CLINICAL TRIAL: NCT01911065
Title: T Cell Responses to Varicella Zoster Virus After Vaccination and Viral Escape
Brief Title: T Cell Responses to Varicella Zoster Virus (VZV) Vaccine SLVP020
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Cornelia L. Dekker, Professor, Pediatrics, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SU-19385; 1U19AI090019-01 (NIH)
Record Dates: First submitted 2013-07-17; First posted 2013-07-30 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-11

CONDITIONS: Herpes Zoster
Keywords: Herpes zoster; immune response; Zostavax; twins; non-twins
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zostavax™ vaccine group (Experimental): Participants > 50 years will receive a single dose 0.65 ml Zostavax™ (live, attenuated zoster vaccine) administered by subcutaneous injection.
  Interventions: Biological: Zostavax™
- Natural-acquired VZV immunity (No Intervention): Participants 40-49 years of age will not receive any intervention with the objective of examining the influence of age and inherited factors on the varicella zoster virus (VZV)-specific immune response in those with a naturally-acquired VZV immunity (a prior history of chicken pox).

INTERVENTIONS:
Biological: Zostavax™ — In the Vaccination arm, healthy individuals will be vaccinated with the licensed zoster vaccine, Zostavax.
  Other Names: Zoster Vaccine Live
  Arms: Zostavax™ vaccine group

SUMMARY:
In this study the investigators are trying to identify immune signatures that are associated with effective or poor vaccine responses to naturally-acquired herpes zoster virus and the zoster (shingles) vaccine, Zostavax.

DETAILED DESCRIPTION:
This study will examine the frequency, phenotype and repertoire of VZV-specific T cells. The frequency and T-Cell Receptor (TCR) diversity of VZV-specific T cells on days 7 and 14 after vaccination will be examined. The titer of anti-VZV antibodies and T cell frequencies will be examined on day 28 post vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy adult non-twins and twin pairs, 40-49 years of age (Cross-Sectional study) or 50 years of age and older (Vaccination study). If a volunteer cannot participate in the Vaccination study after screening, may be considered for Cross-Sectional study.
* History of prior chicken pox infection or living within the continental U.S. for past 30 years
* Willing to complete the informed consent process
* Availability for follow-up for the planned duration of the study (Cross-Sectional study: 1 visit; Vaccination study: 5 visits within 4-5 weeks)
* Acceptable medical history and vital signs

Exclusion Criteria:

* History of shingles within 5 years of enrollment
* Prior vaccination with Zostavax vaccine for prevention of shingles
* Vaccination Study only: History of severe allergic reactions to vaccine components, including gelatin and neomycin.
* Vaccination Study only: Life-threatening reactions to previous vaccinations.
* Vaccination Study only: Adults weighing less than 110 pounds.
* Active systemic or serious concurrent illness, including febrile illness on the day of enrollment/vaccination
* History of immunodeficiency disorder
* Chronic HIV, Hepatitis B or Hepatitis C infection
* Known or suspected impairment of immunologic function, including, but not limited to clinically significant liver disease, diabetes mellitus treated with insulin, moderate to severe renal disease or any other chronic disorder which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
* Recent or current use of immunosuppressive medication, or anticipated use during study period, including systemic corticosteroids (corticosteroid nasal sprays, inhaled steroids and topical steroids are permissible).
* Blood pressure >150 systolic or > 95 diastolic at Visit 1
* History of chemotherapy treatment for cancer.
* Malignancy, other than squamous cell or basal cell skin cancer (includes solid tumors such as breast cancer with recurrence in the past year and any hematologic cancer such as leukemia or lymphoma) which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol. Prostate cancer may be acceptable if no metastases and not undergoing treatment with immunosuppressive medications.
* Autoimmune disease, including rheumatoid arthritis, treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel, which in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol (thyroid disease may be acceptable).
* History of blood dyscrasias, renal disease, or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year
* Use of anti-coagulation medication such as Coumadin or Lovenox, or anti-platelet agents such as aspirin (except aspirin up to 325 mg. daily), Plavix or Aggrenox which may, in the opinion of the investigator, jeopardize volunteer safety or compliance with the protocol.
* Receipt of blood or blood products within 6 months prior to enrollment and during the study period
* Use of antiviral medications within 24 hrs. prior to enrollment, and for the Vaccination study, for the 14 days following study vaccination.
* Inactivated vaccine within 14 days prior to enrollment and during study period(avoid non-study related immunization during the study period)
* Live, attenuated vaccine within 60 days prior to enrollment and during study period (avoid non-study related immunization during the study period)
* Pregnant or lactating woman, planning to become pregnant (pregnancy should be avoided for 3 months following administration of Zostavax vaccine).
* Use of investigational agents within 30 days prior to enrollment and during study period
* Donation of a unit of blood within 6 weeks prior to enrollment and during study period
* Medical or psychiatric condition or occupational responsibilities that preclude subject compliance with the protocol
* Any condition which, in the opinion of the investigator, might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia L Dekker, MD, Principal Investigator — Stanford University; Jorg J Goronzy, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang C, Liu Y, Cavanagh MM, Le Saux S, Qi Q, Roskin KM, Looney TJ, Lee JY, Dixit V, Dekker CL, Swan GE, Goronzy JJ, Boyd SD. B-cell repertoire responses to varicella-zoster vaccination in human identical twins. Proc Natl Acad Sci U S A. 2015 Jan 13;112(2):500-5. doi: 10.1073/pnas.1415875112. Epub 2014 Dec 22. PMID 25535378
- [Background] Fang F, Yu M, Cavanagh MM, Hutter Saunders J, Qi Q, Ye Z, Le Saux S, Sultan W, Turgano E, Dekker CL, Tian L, Weyand CM, Goronzy JJ. Expression of CD39 on Activated T Cells Impairs their Survival in Older Individuals. Cell Rep. 2016 Feb 9;14(5):1218-1231. doi: 10.1016/j.celrep.2016.01.002. Epub 2016 Jan 28. PMID 26832412
- [Background] Qi Q, Cavanagh MM, Le Saux S, NamKoong H, Kim C, Turgano E, Liu Y, Wang C, Mackey S, Swan GE, Dekker CL, Olshen RA, Boyd SD, Weyand CM, Tian L, Goronzy JJ. Diversification of the antigen-specific T cell receptor repertoire after varicella zoster vaccination. Sci Transl Med. 2016 Mar 30;8(332):332ra46. doi: 10.1126/scitranslmed.aaf1725. PMID 27030598
- [Background] Qi Q, Cavanagh MM, Le Saux S, Wagar LE, Mackey S, Hu J, Maecker H, Swan GE, Davis MM, Dekker CL, Tian L, Weyand CM, Goronzy JJ. Defective T Memory Cell Differentiation after Varicella Zoster Vaccination in Older Individuals. PLoS Pathog. 2016 Oct 20;12(10):e1005892. doi: 10.1371/journal.ppat.1005892. eCollection 2016 Oct. PMID 27764254

RESULTS

PARTICIPANT FLOW:
Groups:
- Zostavax™ Vaccine Group: Participants > 50 years received a single dose 0.65 ml Zostavax™ (live, attenuated zoster vaccine) administered by subcutaneous injection.
- Naturally-acquired VZV Immunity: Participants 40-49 years of age did not receive any intervention with the objective of examining the influence of age and inherited factors on the varicella zoster virus (VZV)-specific immune response in those with a naturally-acquired VZV immunity (a prior history of chicken pox).
Period: Overall Study
Arm/Group | Zostavax™ Vaccine Group | Naturally-acquired VZV Immunity
Started | 45 | 9
Completed | 45 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zostavax™ Vaccine Group | Naturally-acquired VZV Immunity | Total
Number analyzed (Participants) | 45 | 9 | 54
Age, Customized [Count of Participants; unit: Participants]
  Age: 40-49 Years Old | 0 | 9 | 9
  Age: 50 and above | 45 | 0 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 7 | 28
  Male | 24 | 2 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 40 | 9 | 49
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 43 | 7 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 45 | 9 | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received Zostavax Immunization or Had Natural Exposure to VZV
Time Frame: Day 0 to Day 35
Measure: Count of Participants; unit: Participants
Arm/Group | Zostavax™ Vaccine Group | Naturally-acquired VZV Immunity
Number analyzed (Participants) | 45 | 9
Participants | 45 | 9

2. Secondary Outcome: Number of Participants With Related Adverse Events
Time Frame: 0 to 35 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Zostavax™ Vaccine Group | Naturally-acquired VZV Immunity
Number analyzed (Participants) | 45 | 9
Participants
  Erythema at injection site greater 5 cm | 5 | 0
  No related AEs | 40 | 9

3. Other Pre Specified Outcome: Identify Predictors That Correlate With a Rapid and Diverse T Cell Response.
Description: The investigators will use the frequency and TCR diversity of VZV-specific T cells on days 7 and 14 after vaccination as outcome variable and identify predictors that positively or negatively correlate with a rapid and diverse T cell response in the different age groups.
Time Frame: 0 to 14 Days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Zostavax™ Vaccine Group | Naturally-acquired VZV Immunity
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/9
Other Adverse Events (participants affected / at risk) | 3/45 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zostavax™ Vaccine Group (N=45) | Naturally-acquired VZV Immunity (N=9)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — Resolved without sequelae
Herpes zoster (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Herpes zoster developed 1 day following immunization; lesion isolate sent to CDC and was wild-type (not vaccine strain), resolved after prolonged PHN despite prompt antiviral treatment. VAERS report filed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No